CLINICAL TRIAL: NCT00839202
Title: Pharmacokinetic (PK) Analysis of a Novel Immunoassay in Hemophilia A
Brief Title: Activity and Content of Factor VIII (FVIII) in Human Plasma: The Assessment of a Novel Immunoassay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of Vermont (Other)
Responsible Party: Principal Investigator, Edward Gomperts, Attending Hematologist, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCI-06-0069-CR002
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hemophilia A
Keywords: factor VIII; hemophilia A; assay
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FVIII immuno-assay (Experimental): The study is not designed as a therapeutic evaluation, but an assessment of clotting factor VIII timed responses after the infusion of specified doses of licensed clotting factor VIII concentrates. The purpose of the study is to measure the levels of infused licensed clotting factor VIII by standard assay techniques and comparing these standard assays with an experimental assay. Measurements of possible co-factors that might impact the results were also carried out.
  Interventions: Other: FVIII immuno-assay

INTERVENTIONS:
Other: FVIII immuno-assay — There is no intervention. This is a study of the differences in assays.

SUMMARY:
A novel immuno-assay is being evaluated for the measurement of Factor VIII. Current procedure measures a rate assay which is subject to much artefact. The hypothesis is that the new assay will give a reading of absolute quantities of FVIII which will provide a more suitable indicator of FVIII content for clotting factor manufacturers, physicians and patients.

DETAILED DESCRIPTION:
Remnant samples collected in a clinical laboratory are assayed with the new procedure and compared with the standard functional activated partial thromboplastin time (APTT) assay. A PK study in seven study subjects with hemophilia A is being carried out using five different commercially licensed factor VIII concentrates and the blood samples drawn for the PK analysis are being measured for FVIII with the novel assay and compared with the standard APTT assay. The concentrates used in the PK studies are also being applied to the two assay systems to determine each product's specific activity.

ELIGIBILITY:
Inclusion Criteria:

* adults with hemophilia A
* factor VIII less that 2%
* informed consent signed
* absence of an inhibitor

Exclusion Criteria:

* history of a high responding inhibitor anemia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The level of Factor VIII in pMols | 48 hours

SECONDARY OUTCOMES:
The possible role of VWF, factor concentrate type and non-inhibitory antibody presence or absence on the FVIII antigen levels | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Edward D Gomperts, MD, Principal Investigator — Children's Hospital Los Angeles; Kenneth G Mann, PhD, Principal Investigator — University of Vermont
Locations (1):
- Department of Biochemistry University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No